CLINICAL TRIAL: NCT02433769
Title: Acceleromyographic Assessment of Neuromuscular Blockade: TOF-Watch-SX Versus TOFscan
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn S. Murphy, MD, Director Clinical Research, Endeavor Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EH14-266
Record Dates: First submitted 2015-04-23; First posted 2015-05-05 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Neuromuscular Blockade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TOf-Watch-SX (Active Comparator): Train-of-four (TOF) ratios will be measured with the TOF-Watch-SX and compared to TOF ratios measured simultaneously with the TOFscan
  Interventions: Device: TOF-Watch-SX
- TOFscan (Experimental): Train-of-four (TOF) ratios obtained from the TOFscan will be compared to TOF ratios measured simultaneously with the TOF-Watch-SX
  Interventions: Device: TOFscan

INTERVENTIONS:
Device: TOFscan — Data from the TOFscan will be compared to simultaneously measured data from the TOF-Watch-SX ("gold standard")
  Arms: TOFscan
Device: TOF-Watch-SX — Data from the TOF-Watch-SX will be compared to simultaneously measured data from the TOFscan
  Arms: TOf-Watch-SX

SUMMARY:
Muscle relaxants are administered to most patients undergoing general anesthesia in order to facilitate the placement of an endotracheal tube and improve operating conditions. Despite routine reversal of these agents, many patients arrive in the recovery room with evidence of residual muscle weakness. Many studies have demonstrated that residual neuromuscular blockade (weakness) is a common occurrence after surgery. The only method of reliably detecting the presence of perioperative neuromuscular blockade is through the use of quantitative neuromuscular monitors. These devices measure and quantify the degree of muscle weakness and display the results on a screen. When using train-of-four (TOF) nerve stimulation, the ratio of the fourth muscle contraction (twitch) to the first twitch will be displayed; when this ratio is 90% (or 0.9) or greater, full recovery of muscle strength is present, and the endotracheal tube can be safely removed. At the present time, there is only one commercially-available stand-alone quantitative monitor available in the United States -the TOF-Watch (an acceleromyography device). It is not used by many clinicians because it requires experience to obtain accurate results, is expensive, and is subject to interference by factors in the operating room. The aim of this investigation is to examine a new quantitative monitor, the TOFscan (a new three dimensional acceleromyography device). In order to study the accuracy of this new device, the TOFscan will be compared to the current "clinical gold standard", the TOF-Watch-SX.

DETAILED DESCRIPTION:
30 patients presenting for elective surgical procedures with an expected duration greater than 60 minutes will be enrolled in this study. ASA I to III patients requiring neuromuscular blockade in the operating room will be eligible for enrollment. All neuromuscular management will be conducted as recommended by the Good Clinical Research Practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents guidelines

Monitoring will consist of standard ASA monitors, which include manual blood pressure measurements, continuous EKG monitoring, pulse oximetry, capnography, and infrared gas analysis. The placement of the TOFscan to the dominant or non-dominant hand will be determined using a computer-generated randomization table. The TOF-Watch-SX will be placed on the other hand.

Anesthetic induction will be as per usual routine clinical care, consisting of propofol 2.0-2.5 mg/kg and fentanyl 100 μg; rocuronium 0.6 mg/kg will be given over 5 seconds through a fast-running IV after baseline neuromuscular data are collected. General anesthesia will be maintained with sevoflurane 1.0-3.0%, with the concentration of inhalational agent adjusted to maintain blood pressure within 20% of baseline values. The depth of anesthesia will also be adjusted to maintain Bispectral Index (BIS monitor) values between 40-60, as per usual clinical practice. Core temperature will be maintained > 35°C and hand temperature > 32°C using an upper extremity warming blanket. Additional doses of rocuronium can be administered (5-10 mg) if required for surgical relaxation (a TOF count of 2-3 during TOF stimulation). No NMBAs will be administered during the last 20 minutes of the procedure. At the completion of surgery, neuromuscular blockade will be reversed with neostigmine 50 µg/kg plus glycopyrrolate, per usual standard of care.

Upon arrival to the operating room, neuromuscular monitoring surface electrodes will be applied. All monitoring will be conducted while the patient is under general anesthesia for the surgical procedure. Surface electrodes (non-invasive EKG electrodes) will be placed on the cleansed skin over the ulnar nerve of both arms near the wrist. The electrodes will be connected by leads to the nerve stimulator component of the TOF-Watch-SX on one arm and the TOFscan on the other arm. The transducer (AMG sensor which measures acceleration) of the TOF-Watch-SX will be placed on the thumb of the corresponding hand. A 75-150g preload (via the Hand adapter) will be applied as per standard recommendations. On the other hand, the transducer (three-dimensional AMG sensor) of the TOFscan will be placed on the thumb using the integrated hand adapter. During the surgical procedure, both devices will be activated simultaneously, and the responses to nerve stimulation recorded.

After induction of anesthesia, but before administration of rocuronium, calibration and stable baseline signals will be achieved for the TOF-Watch-SX and the TOFscan as suggested by the Good Clinical Research Guidelines. After the baseline data are collected, the neuromuscular blocking agent (rocuronium) will be administered. Data relating to onset (a TOF ratio decreases from 1.0 to 0.3 or less on the TOF-Watch-SX display), maintenance (the TOF ratio is less than 0.3 and constant on the TOF-Watch-SX display), and reversal (an increase in the TOF ratio from 0.2 to 0.9 or above) will be recorded. At these same times, data from the TOFscan will be recorded. Monitoring will continue until full recovery of neuromuscular function is noted (a TOF ratio of at least 0.9 or greater on the TOF-Watch-SX device display). At this time, the anesthesia agents will be turned off and the patient awakened and extubated. After surgery, data recorded simultaneously from the TOF-Watch-SX and the TOFscan will be compared.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III patients requiring neuromuscular blockade in the operating room

Exclusion Criteria:

* presence of an underlying neuromuscular disease
* use of drugs known to interfere with neuromuscular transmission (antiseizure medications, anticholinesterases, magnesium sulfate)
* presence of renal or hepatic disease
* procedures preventing access to both of the upper extremities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Train-of-four (TOF) ratio 0.7 | from the start of surgery until 1 hour after admission to the recovery room
  Data from the TOFscan will be compared to the TOF-Watch-SX at a TOF ratio of 0.7 (when the TOF-Watch-SX reads 0.7 (gold standard), the reading from the TOFscan will be recorded and compared

SECONDARY OUTCOMES:
Train-of-four (TOF) ratio 0.6 | from the start of surgery until 1 hour after admission to the recovery room
  Data from the TOFscan will be compared to the TOF-Watch-SX at a TOF ratio of 0.6 (when the TOF-Watch-SX reads 0.6 (gold standard), the reading from the TOFscan will be recorded and compared
train-of-four (TOF) ratio 0.9 | from the start of surgery until 1 hour after admission to the recovery room
  Data from the TOFscan will be compared to the TOF-Watch-SX at a TOF ratio of 0.9 (when the TOF-Watch-SX reads 0.9 (gold standard), the reading from the TOFscan will be recorded and compared

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States